CLINICAL TRIAL: NCT02552511
Title: A Multi-Centre Epidemiology Study on Neonatal Seizure in China
Brief Title: Epidemiology Study on Neonatal Seizure
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: Xiamen Children's Hospital, Fujian of China (Other); Maternal and Child Health Hospital of Guangxi Zhuang Autonomous Region (Other); Guangzhou Women and Children's Medical Center (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Maternal and Child Health Hospital of Hubei Province (Other); The People's Hospital of Dehong Autonomous Prefecture (Other); Guangzhou Medical University (Other); Nanfang Hospital of Southern Medical University, Guangdong of China (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHFudanU_NNICU6; NCT02605031 (obsolete NCT alias)
Record Dates: First submitted 2015-09-04; First posted 2015-09-17 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Exposure: Perinatal factors exposure

SUMMARY:
A Multicentre, observational and cohort study to get the incidence of new-onset or newly-diagnosed seizure in neonatal population. EEG will used to record the change of brain electric activity and diagnose. Other data also will be collected since first seizure until confirmed diagnosis.

DETAILED DESCRIPTION:
This study is designed to describe the incidence of newborn with uncontrolled seizures. Seizures can be associated with any high-risk factors during perinatal stage and diagnosed by abnormal electrical activity in the brain.

In this study researchers will use electroencephalography (EEG) to determine and monitor newborn with uncontrolled or suspected seizures. EEG works by measuring electrical activity in different areas of the brain. The EEG allows researchers to examine changes in the EEG along with the clinical features of seizures as they occur.

In addition to monitoring electrical activity of the brain, researchers will collect demographic, medical history, family, perinatal stage, birth, growth, feeding condition by medical records and questionnaire. These information will allow researchers to learn more about what high-risk factors influence the incidence of neonatal seizure in China.

ELIGIBILITY:
Inclusion Criteria:

* Age from 0~28 days;
* Clinical diagnosed with seizure;
* EEG diagnosed with seizure;
* Parents who consent to their participation in the study;

Exclusion Criteria:

* Parents who will not comply to the needs and the design process.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All inpatients and Outpatients of neonates
Sampling Method: Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of new-onset or newly-diagnosed seizure in the neonatal population and stratified by epilepsy status. | Participants will be followed for the duration of neonatal from birth to 28 day, an expected average of 28 days.
  Incidence of new-onset or newly-diagnosed seizure in the neonatal population and stratified by epilepsy status.

SECONDARY OUTCOMES:
EEG | In 14 Days after seizure attack
  To measured by EEG after seizure attack.
Neurodevelopment(Bayley Scores) | At corrected age of 18 months
  To evaluate neurodevelopmental function via Bayley Scores of Infant Development Mental Development Index (BSID) and gain incidence of MDI<70(Severe) or MDI<85(Moderate).
Neurological Evaluation(GMFM-88 Scores) | At corrected age of 18 months
  To gain changes in standardized gross motor function using GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales, lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 , Higher value means better gross motor function).malformation using genomic methods.
Gene Mutation | 30 days after receipt of DNA sample
  To detect the mutation and characterize the genetic architecture and risk variants of neonatal malformation using genomic methods.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhao Zhou, Doctor, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Sen S, Keough K, Gibson J. Clinical reasoning: novel GLUT1-DS mutation: refractory seizures and ataxia. Neurology. 2015 Apr 14;84(15):e111-4. doi: 10.1212/WNL.0000000000001467. PMID 25870456
- [Background] Lateef TM, Johann-Liang R, Kaulas H, Hasan R, Williams K, Caserta V, Nelson KB. Seizures, encephalopathy, and vaccines: experience in the National Vaccine Injury Compensation Program. J Pediatr. 2015 Mar;166(3):576-81. doi: 10.1016/j.jpeds.2014.10.054. Epub 2014 Dec 2. PMID 25477158
- [Background] Payne ET, Zhao XY, Frndova H, McBain K, Sharma R, Hutchison JS, Hahn CD. Seizure burden is independently associated with short term outcome in critically ill children. Brain. 2014 May;137(Pt 5):1429-38. doi: 10.1093/brain/awu042. Epub 2014 Mar 4. PMID 24595203
- [Background] Sanchez Fernandez I, Abend NS, Arndt DH, Carpenter JL, Chapman KE, Cornett KM, Dlugos DJ, Gallentine WB, Giza CC, Goldstein JL, Hahn CD, Lerner JT, Matsumoto JH, McBain K, Nash KB, Payne E, Sanchez SM, Williams K, Loddenkemper T. Electrographic seizures after convulsive status epilepticus in children and young adults: a retrospective multicenter study. J Pediatr. 2014 Feb;164(2):339-46.e1-2. doi: 10.1016/j.jpeds.2013.09.032. Epub 2013 Oct 22. PMID 24161223
- [Background] Iyer A, Appleton R. Management of reflex anoxic seizures in children. Arch Dis Child. 2013 Sep;98(9):714-7. doi: 10.1136/archdischild-2012-303133. Epub 2013 Jun 28. PMID 23814085
- [Background] Grunebaum A, McCullough LB, Sapra KJ, Brent RL, Levene MI, Arabin B, Chervenak FA. Apgar score of 0 at 5 minutes and neonatal seizures or serious neurologic dysfunction in relation to birth setting. Am J Obstet Gynecol. 2013 Oct;209(4):323.e1-6. doi: 10.1016/j.ajog.2013.06.025. Epub 2013 Jun 19. PMID 23791692
- [Background] Beslow LA, Abend NS, Gindville MC, Bastian RA, Licht DJ, Smith SE, Hillis AE, Ichord RN, Jordan LC. Pediatric intracerebral hemorrhage: acute symptomatic seizures and epilepsy. JAMA Neurol. 2013 Apr;70(4):448-54. doi: 10.1001/jamaneurol.2013.1033. PMID 23392319
- [Background] Kidokoro H, Kubota T, Hayakawa M, Kato Y, Okumura A. Neonatal seizure identification on reduced channel EEG. Arch Dis Child Fetal Neonatal Ed. 2013 Jul;98(4):F359-61. doi: 10.1136/archdischild-2012-302361. Epub 2012 Oct 27. PMID 23104986
- [Background] Wilden JA, Cohen-Gadol AA. Evaluation of first nonfebrile seizures. Am Fam Physician. 2012 Aug 15;86(4):334-40. PMID 22963022